CLINICAL TRIAL: NCT05318729
Title: Application of a Unique Vibration Modality for Postoperative Pain Control in Patients With Distal Radius Fractures to Reduce Postoperative Pain and Opioid Use
Brief Title: Use of a Vibration Tool for Postoperative Pain Control in Distal Radius Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jason Ko, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00214664
Record Dates: First submitted 2022-03-08; First posted 2022-04-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Distal Radius Fracture; Radius Fracture Distal; Radius; Fracture, Lower or Distal End; Postoperative Pain
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vibration tool (Experimental): Use of the vibration tool 3 times per day for 10 minutes for each session Morning, mid-day, and evening.
  Volarly for 5 minutes and dorsally for 5 minutes, for a total of 10 minutes during each session:
  Interventions: Device: Vibration tool
- Control (No Intervention): Standard of care, no vibration tool.

INTERVENTIONS:
Device: Vibration tool — Therapeutic mini massager for scar management, desensitization, muscle stimulation, oral stimulation and sensory re-education. Seek pain relief for sore achy muscles, tendons or bones.
  Other Names: Norco NC70209 Mini Massager
  Arms: Vibration tool

SUMMARY:
The purpose of this research study is to determine if using a vibration tool improves pain control after surgical treatment of distal radius fracture. Additionally, the investigators would like to determine if this tool has any impact on consumption of pain medications postoperatively.

DETAILED DESCRIPTION:
Traditionally, occupational therapists have utilized vibration for sensory re-education in compression neuropathies and peripheral nerve injuries. Vibration is also commonly used for desensitization of hypersensitivity following amputation, crush injury, and for hypersensitive scarring. Since the vibration tool is readily available in the hand therapy clinic, vibration analgesia should be further explored in the hand clinic to help reduce pain. Vibration is a simple, and non-invasive, tool and would be easy, economical, and practical to implement into the hand clinic for postoperative pain control. This research project will evaluate whether vibration can be a useful adjunct to current postoperative pain modalities. With a multidisciplinary approach, the investigators hope to highlight the use of non-opioid modalities of pain control in distal radius fractures and believe that the findings from this study may apply to other painful conditions of the hand as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a distal radius fracture who have undergone an open reduction and internal fixation using a volar FCR approach with a single volar plate
* Patients who can read, write, and follow direction in English
* Willing to undergo occupational therapy at Northwestern Medicine's Hand Surgery clinic

Exclusion Criteria:

* Patients undergoing oncologic surgery
* Patients who undergo simultaneous surgery such as open carpal tunnel
* Patients who only require closed reduction of distal radius fractures
* Operative patients that require dorsal plate fixation or separate radial styloid plate fixation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
QuickDASH (Disabilities of the Arm, Shoulder, and Hand) Questionnaire | up to 8 week post-surgery
  An 11-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb; scored from 0 (no disability) to 100 (most severe disability).
PROMIS Bank v1.1 - Pain Interference Computer Adaptive Test | up to 8 weeks post-surgery
  A 4-6 item self-reported questionnaire designed to measure the consequences of pain on relevant aspects of a person's life; the T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10; low scores represent less pain interference, while high scores represent greater interference.
PROMIS Bank v2.0 - Upper Extremity Computer Adaptive Test | up to 8 weeks post-surgery
  A 4-6 item self-reported questionnaire designed to measure upper extremity function; the T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10; low scores represent less function, while high scores represent greater function.
Pain Visual Analog Scale (VAS) | up to 8 weeks post-surgery
  Scored from 0 (no pain) to 10 (worst possible pain)

SECONDARY OUTCOMES:
Opioid Use | up to 8 weeks post-surgery
  Number of opioid pain medication tablets consumed

CONTACTS AND LOCATIONS:
Overall Officials: Jason H Ko, MD, MBA, Principal Investigator — Associate Professor
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No